CLINICAL TRIAL: NCT03399175
Title: Influência de imunomodulação Precoce Influence of Early Immunosuppressive Therapy on the Course of Vogt-Koyanagi-Harada Disease: a Prospective Study
Brief Title: Early Immunosuppressive Therapy on the Course of Vogt-Koyanagi-Harada Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Joyce Hisae Yamamoto, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VKH Brazilian Study Group
Record Dates: First submitted 2017-11-26; First posted 2018-01-16 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Vogt Koyanagi Harada Disease
Keywords: Vogt-Koyanagi-Harada disease; Immunosuppressive therapy; Indocyanine green angiography; Enhanced depth imaging optical coherence tomography; Electroretinogram
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome | interventions — Adrenal Cortex Hormones; Immunosuppression Therapy

STUDY DESIGN:
Intervention Model Description: Early systemic high-dose corticosteroid and immunosuppressive therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Other): Early high-dose corticosteroid and immunosuppressive therapy
  Interventions: Drug: Early high-dose corticosteroid and immunosuppressive therapy

INTERVENTIONS:
Drug: Early high-dose corticosteroid and immunosuppressive therapy — Early high-dose corticosteroid and immunosuppressive therapy
  Other Names: Treatment group

SUMMARY:
This prospective study will include patients with Vogt-Koyanagi-Harada disease from disease onset, treated with early systemic high-dose corticosteroid and immunosuppressive therapy. Clinical and subclinical signs of disease activity added with electroretinogram exams, through predefined intervals, will be evaluated through a minimum 12-month follow-up.

DETAILED DESCRIPTION:
Vogt-Koyanagi-Harada disease (DVKH) is an autoimmune disorder, which is mainly a T CD4+ Th1 lymphocyte mediated aggression to melanocytes, in individuals with a genetic predisposition, in particular, the presence of HLA-DRB1*0405 allele. It is an important cause of non-infectious uveitis at tertiary services in Brazil and a major cause of uveitis in general, in some regions of the world, such as in Japan and Asia. Its clinical course is classically defined in four phases: prodromal, with general symptoms possibly related to a viral trigger; uveitic, with sudden decrease in visual acuity in both eyes with a diffuse choroiditis associated or not to iridocyclitis; convalescent, wherein the depigmentation of the integument and choroid is more evident, with an apparently quiescent disease from a clinical point of view; and chronic or recurrent, in which the predominant inflammatory signs of anterior segment are clinically detected and complications are more evident, such as choroidal neovascularization, cataract and glaucoma.

Recent studies have shown subclinical inflammation of the choroid, detected by indocyanine green angiography (ICGA) and also by enhanced-depth imaging spectral-domain optical coherence tomography (EDI-OCT). Several authors have been taking these findings into account for inflammation monitoring and treatment follow-up. However, the wider knowledge of these subclinical signs of inflammation and the understanding of the disease's course from a global perspective are still scarce. The study developed by Sakata et al. (2012-2015) established an early and aggressive treatment with pulsetherapy of methylprednisolone, followed by high doses of oral prednisone (1 mg / kg / day) with slow and gradual tapering over a 15-month period. Such study has showed that, despite an "adequate" treatment: a) 94% of patients had worsening of visual acuity or disease relapse during a 12-month follow-up; b) subclinical signs fluctuated without changing the initial treatment ; c) particular cases, in which there was an increase of treatment, showed better retinal function at final follow-up.

Thus, this study aims to continue the evaluation of subclinical signs and their clinical and functional relevance, as well as, with an early immunomodulatory treatment, to observe the clinical course of DVKH and its behavior in functional terms and development of complications. Study design: prospective and longitudinal, with a minimum 12-month follow-up, with integrated clinical, angiographic, tomographic and functional assessments. On clinical examination, anterior segment inflammatory signs will be evaluated (cells in anterior chamber), as well as posterior findings (observed in the acute phase: optic disc hyperemia, exudative retinal detachment, macular edema, vasculitis, vitreous haze); on angiographic evaluation, fluorescein angiogram (FA) and ICGA will be included; on tomographic evaluation, evaluation of retina and choroid will be included (EDI-OCT); and, on the functional tests, it will be included: the full-field electroretinography (ERGct) and multifocal electroretinography (ERGmf); as well as autofluorescence (AF) with blue light (Bl-AF) and near-infrared light (NIR-AF); automated perimetry (30-2) and contrast sensitivity test. Quality of life questionnaires and visual function evaluation will be included in pre-defined intervals.

Expected results: 1. To reaffirm the importance of an integrated analysis of the clinical and ancillary tests for better patient monitoring and to improve disease prognosis; 2. To increase the understanding of the disease natural course; 3. To increase the understanding of the disease pathogenesis; and, 4. To set parameters (outcomes) that can guide therapy.

ELIGIBILITY:
Inclusion criteria:

- acute Vogt-Koyanagi-Harada disease

Exclusion criteria:

* non collaborative patient
* minimum one-year follow-up

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03-23 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
scotopic electroretinogram results | 6 month; 12 month
  scotopic results variation between 12 months and 6 months

SECONDARY OUTCOMES:
presence of optic disc hyperfluorescence detected on fluorescein angiography | between 6 and 12 months from disease onset.
  presence of optic disc hyperfluorescence and variation in intensity in consecutive examinations
presence of perivascular leakage on fluorescein angiography | between 6 and 12 months from disease onset.
  presence of perivascular leakage and variation in extension and intensity in consecutive examinations
presence of dark dots on indocyanine green angiography | between 6 and 12 months from disease onset.
  dark dots score and its fluctuation
subfoveal choroidal thickness on enhanced depth imaging optical coherence tomography | between 6 and 12 months from disease onset.
  subfoveal choroidal thickness and its variation
presence of cells in anterior chamber graduated according to SUN criteria | between 6 and 12 months from disease onset.
  presence of cells in anterior chamber and its variation
presence of choroidal neovascular membrane on OCT and/or FA | between 6 and 12 months from disease onset.
  choroidal neovascular membrane
presence of macular edema on OCT and/or FA | between 6 and 12 months from disease onset.
  macular edema detected clinically, angiographically and/or by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Joyce H Yamamoto, MD, Principal Investigator — University of Sao Paulo School of Medicine Ophthalmology
Locations (1):
- Hospital das Clinicas HCFMUSP, Faculdade de Medicina Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lavezzo MM, Sakata VM, Morita C, Rodriguez EE, Abdallah SF, da Silva FT, Hirata CE, Yamamoto JH. Vogt-Koyanagi-Harada disease: review of a rare autoimmune disease targeting antigens of melanocytes. Orphanet J Rare Dis. 2016 Mar 24;11:29. doi: 10.1186/s13023-016-0412-4. PMID 27008848
- [Result] Sakata VM, da Silva FT, Hirata CE, de Carvalho JF, Yamamoto JH. Diagnosis and classification of Vogt-Koyanagi-Harada disease. Autoimmun Rev. 2014 Apr-May;13(4-5):550-5. doi: 10.1016/j.autrev.2014.01.023. Epub 2014 Jan 15. PMID 24440284
- [Result] Damico FM, Bezerra FT, Silva GC, Gasparin F, Yamamoto JH. New insights into Vogt-Koyanagi-Harada disease. Arq Bras Oftalmol. 2009 May-Jun;72(3):413-20. doi: 10.1590/s0004-27492009000300028. PMID 19668980
- [Result] da Silva FT, Damico FM, Marin ML, Goldberg AC, Hirata CE, Takiuti PH, Olivalves E, Yamamoto JH. Revised diagnostic criteria for vogt-koyanagi-harada disease: considerations on the different disease categories. Am J Ophthalmol. 2009 Feb;147(2):339-345.e5. doi: 10.1016/j.ajo.2008.08.034. Epub 2008 Nov 7. PMID 18992868
- [Result] da Silva FT, Hirata CE, Olivalves E, Oyamada MK, Yamamoto JH. Fundus-based and electroretinographic strategies for stratification of late-stage Vogt-Koyanagi-Harada disease patients. Am J Ophthalmol. 2009 Dec;148(6):939-45.e3. doi: 10.1016/j.ajo.2009.06.029. Epub 2009 Sep 24. PMID 19781687
- [Result] da Silva FT, Hirata CE, Sakata VM, Olivalves E, Preti R, Pimentel SL, Gomes A, Takahashi WY, Costa RA, Yamamoto JH. Indocyanine green angiography findings in patients with long-standing Vogt-Koyanagi-Harada disease: a cross-sectional study. BMC Ophthalmol. 2012 Aug 13;12:40. doi: 10.1186/1471-2415-12-40. PMID 22889440
- [Result] da Silva FT, Sakata VM, Nakashima A, Hirata CE, Olivalves E, Takahashi WY, Costa RA, Yamamoto JH. Enhanced depth imaging optical coherence tomography in long-standing Vogt-Koyanagi-Harada disease. Br J Ophthalmol. 2013 Jan;97(1):70-4. doi: 10.1136/bjophthalmol-2012-302089. Epub 2012 Oct 25. PMID 23099292
- [Result] Sakata VM, da Silva FT, Hirata CE, Takahashi WY, Costa RA, Yamamoto JH. Choroidal bulging in patients with Vogt-Koyanagi-Harada disease in the non-acute uveitic stage. J Ophthalmic Inflamm Infect. 2014 Feb 18;4(1):6. doi: 10.1186/1869-5760-4-6. PMID 24548697
- [Result] Sakata VM, da Silva FT, Hirata CE, Marin ML, Rodrigues H, Kalil J, Costa RA, Yamamoto JH. High rate of clinical recurrence in patients with Vogt-Koyanagi-Harada disease treated with early high-dose corticosteroids. Graefes Arch Clin Exp Ophthalmol. 2015 May;253(5):785-90. doi: 10.1007/s00417-014-2904-z. Epub 2015 Jan 16. PMID 25592477
- [Result] Morita C, Sakata VM, Rodriguez EE, Abdallah SF, Lavezzo MM, da Silva FT, Machado CG, Oyamada MK, Hirata CE, Yamamoto JH. Fundus autofluorescence as a marker of disease severity in Vogt-Koyanagi-Harada disease. Acta Ophthalmol. 2016 Dec;94(8):e820-e821. doi: 10.1111/aos.13147. Epub 2016 Jul 2. No abstract available. PMID 27368955
- [Result] Herbort CP Jr, Abu El Asrar AM, Yamamoto JH, Pavesio CE, Gupta V, Khairallah M, Tugal-Tutkun I, Soheilian M, Takeuchi M, Papadia M. Reappraisal of the management of Vogt-Koyanagi-Harada disease: sunset glow fundus is no more a fatality. Int Ophthalmol. 2017 Dec;37(6):1383-1395. doi: 10.1007/s10792-016-0395-0. Epub 2016 Nov 14. PMID 27844182